CLINICAL TRIAL: NCT04805476
Title: Prophylactic Use of Noninvasive Ventilation in the Postoperative Period of Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 50468415.1.0000.5327
Record Dates: First submitted 2020-11-03; First posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Bariatric Surgery Candidate; Obesity, Morbid; Ventilatory Failure
MeSH Terms: conditions — Obesity, Morbid; Hypoventilation | interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non invasive mechanical ventilation (Experimental): The subjects in the immediate intervention group (GI) will be extubated and placed in NIV the moment they enter the recovery room through a portable ventilator (Esprit ® or BiPAP Vision ®, Respironics) in face mask. The parameters will be adjusted as follows: FiO2 = 50%, positive expiratory pressure (EPAP, starting at 4-6 cmH2O and adjusting 1-2 cmH2O to avoid snoring, apnea, paradoxical breathing and desaturations) and adjusted inspiratory positive pressure (IPAP) to maintain a tidal volume of 400 to 500 ml, maintaining IPAP <15cmH2O17. Individuals will receive this ventilatory support for 1 hour. After this period the patients will be submitted to the same care of GP patients.
  Interventions: Device: Non invasive mechanical ventilation
- Usual care (Active Comparator): Subjects will receive oxygen therapy through a nasal cannula with 4 to 6 L / min of oxygen according to the team routine and patient need.
  Interventions: Device: GP

INTERVENTIONS:
Device: Non invasive mechanical ventilation — Prophylactic non invasive mechanical ventilation
  Arms: Non invasive mechanical ventilation
Device: GP — GP subjects will receive oxygen therapy through a nasal cannula with 4 to 6 L / min of oxygen according to team routine and patient need.
  Arms: Usual care

SUMMARY:
Comorbidities associated with severe obesity determine an important public health problem. Few methods are considered potentially effective for the treatment of severe obesity and the clinical relevance of bariatric surgery is growing, as well as the number of procedures performed. The insertion of the physiotherapist in the multiprofessional team responsible for performing the surgical procedure is essential from the preoperative screening and evaluation to the prevention and treatment of postoperative complications. Therefore, the physiopathological aspects involved with severe obesity, the technical aspects and risks of the surgical procedure, as well as the physiotherapeutic techniques that have scientific proof must be known by the physiotherapist responsible for the surgical follow-up of the patient. In this context, the use of non-invasive ventilation (NIV) in the postoperative period of bariatric surgery has ample therapeutic potential. The present research project aims to evaluate the immediate prophylactic use of NIV on the respiratory and functional recovery of the patients.

DETAILED DESCRIPTION:
The study will be performed at the surgical center of the Hospital de Clínicas of Porto Alegre. After approval by the Research Ethics Committee, patients must sign the Term of Consent for inclusion in the study. A blinded investigator will record clinical, anthropometric, pulmonary function tests, and functional measures. Patients submitted to open bariatric surgery will be divided into two groups for the use of NIV: immediate post-extubation (IG) and non-intervention (standard group [GP]). Patients will be randomly assigned to the groups. All subjects will undergo general anesthesia and postoperative analgesia, using a standardized surgical team approach. Patients who present the contraindication criteria for the use of NIV will be excluded from the study.

After the surgical procedure and extubation, GP subjects will receive oxygen therapy through a nasal cannula with 4 to 6 L / min of oxygen according to the team routine and patient need. The subjects in the immediate intervention group (GI) will be extubated and placed in NIV the moment they enter the recovery room through a portable ventilator (Esprit ® or BiPAP Vision ®, Respironics) in face mask. The parameters will be adjusted as follows: FiO2 = 50%, positive expiratory pressure (EPAP, starting at 4-6 cmH2O and adjusting 1-2 cmH2O to avoid snoring, apnea, paradoxical breathing and desaturations) and adjusted inspiratory positive pressure (IPAP) to maintain a tidal volume of 400 to 500 ml, maintaining IPAP <15cmH2O17. Individuals will receive this ventilatory support for 1 hour. After this period the patients will be submitted to the same care of GP patients. Measurement of respiratory muscle strength and lung function will be recorded in Time 1 (in the preoperative period), Time 2 (at the time of entry of the recovery room) and Time 3 (1 hour after extubation, with withdrawal of the support ventilatory). Vital signs (heart rate, peripheral O2 Saturation and Blood Pressure) will also be recorded through the multi-parameter monitor (IntelliVue MP40).

The functional evaluation will be performed in the period of the initial data collection through the Functional Status Score for the ICU (FSS-ICU) and Functional Independence Measure (MIF). Patients will be monitored during the hospitalization period until hospital discharge and records of postoperative complications (radiological changes, infections and surgical anastomosis fistulas) will be recorded by blinded evaluator. The final evaluation will be done through the MIF, through telephone contact 1 month after the surgery.

During the study participation patients may present with discomfort, nausea, vomiting and / or pain related to the use of non-invasive ventilation and procedures performed to evaluate muscle strength, lung function and functionality. In a study with methodology and similar population, such risks / complications were not reported16, however, if they occur, the procedures will be immediately interrupted and patients will be assisted by the study researchers in order to preserve the patients and the reliability of the results.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing bariatric surgery

Exclusion Criteria:

* Absolute or relative contraindications to the use of NIV

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) | Preoperative
  Larger volume of air mobilized on an exhalation.
Forced Vital Capacity (FVC) | 10 minutes after admission to the recovery room
  Larger volume of air mobilized on an exhalation.
Forced Vital Capacity (FVC) | 1 hour after admission to the recovery room
  Larger volume of air mobilized on an exhalation.
Forced expiratory volume in one second (FEV1) | Preoperative
  Volume of air exhaled in the first second during the FVC maneuver.
Forced expiratory volume in one second (FEV1) | 10 minutes after admission to the recovery room
  Volume of air exhaled in the first second during the FVC maneuver.
Forced expiratory volume in one second (FEV1) | 1 hour after admission to the recovery room
  Volume of air exhaled in the first second during the FVC maneuver.
FEV1/FVC ratio | Preoperative
  Ratio between forced expiratory volume in the first second and vital capacity.
FEV1/FVC ratio | 10 minutes after admission to the recovery room
  Ratio between forced expiratory volume in the first second and vital capacity.
FEV1/FVC ratio | 1 hour after admission to the recovery room
  Ratio between forced expiratory volume in the first second and vital capacity.
Peak expiratory flow (PEF) | Preoperative
  Maximum air flow during the FVC maneuver.
Peak expiratory flow (PEF) | 10 minutes after admission to the recovery room
  Maximum air flow during the FVC maneuver.
Peak expiratory flow (PEF) | 1 hour after admission to the recovery room
  Maximum air flow during the FVC maneuver.

CONTACTS AND LOCATIONS:
Overall Officials: Fábio Di Naso, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No